CLINICAL TRIAL: NCT03576456
Title: Sedative Premedication in Coronary Angiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Wilgenhof Adriaan, Medical Doctor, Principal Investigator, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: awxg2018
Record Dates: First submitted 2018-06-18; First posted 2018-07-03 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Coronary Angiography; Sedative Premedication
Keywords: coronary angiography; premedication; pain; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Intervention Model Description: placebo controlled, double blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alprazolam (Active Comparator): Patients receive alprazolam 0.5 mg 1 hour prior to coronary angiography.
  Interventions: Drug: Alprazolam 0.5 mg
- Placebo Oral Tablet (Placebo Comparator): Patients receive placebo 1 hour prior to coronary angiography.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Alprazolam 0.5 mg — receive alprazolam prior to angio
  Arms: Alprazolam
Drug: Placebo Oral Tablet — receive placebo prior to angio
  Arms: Placebo Oral Tablet

SUMMARY:
Evaluation of the possible positive effect of sedative premedication prior to coronary angiography in regards to pain and anxiety.

DETAILED DESCRIPTION:
Coronary angiography is an invasive procedure that can cause patient discomfort. Sedative premedication before coronary angiography could be used to reduce anxiety and pain, but evidence is lacking. Previous trials were predominantly conducted in men and in coronary interventions with femoral access. Recently, radial access has become the preferred route for performing coronary angiograms (RIVAL trial) In this setting, sedative premedication could be of interest to reduce radial spasms, patient anxiety and pain.

ELIGIBILITY:
Inclusion Criteria:

* elective coronary angiography

Exclusion Criteria:

* planned PCI
* use of sedative medication at home
* use of alcohol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
preprocedural anxiety: visual analogue scale | Assessed before the coronary angiography
  anxiety prior to coronary angiography. Assessed before the procedure through a visual analogue scale for anxiety (VAS-A). The VAS is a visual scale ranging from 0 to 100 with 0 begin no anxiety at all and 100 begin extreme anxiety.
periprocedural pain: visual analogue scale | Assessed after the coronary angiography, within 4 hours.
  pain during to coronary angiography. Assessed after the procedure through a visual analogue scale for pain. The VAS scale is a visual scale ranging from 0 (no pain) to 100 (extreme pain).

SECONDARY OUTCOMES:
radial spasm | during procedure
  spasm of the radial artery as experienced by operator. There is no precise measurement up until today.
vascular site access complication | during procedure
  need to switch to femoral access, assessed by the operator.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Schoors, MD PhD, Study Director — Head of service
Locations (1):
- Adriaan Wilgenhof, Brussels, Jette, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: within 1 month, during 1 year
Access Criteria: researcher